CLINICAL TRIAL: NCT00002030
Title: An Open Label Study to Evaluate the Long-Term Safety and Effectiveness of Aerosol Pentamidine in the Prophylaxis of Pneumocystis Carinii Pneumonia in AIDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisons (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 022E; 87-72B; 88-21
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-11

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Pentamidine; Aerosols; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Pentamidine

INTERVENTIONS:
Drug: Pentamidine isethionate

SUMMARY:
To evaluate the safety, tolerability, and efficacy of long term, bi-weekly administration of aerosol pentamidine when used as a prophylactic agent in patients who have had at least two or more episodes of AIDS-associated Pneumocystis carinii pneumonia (PCP).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT).
* Standard or experimental treatments for an opportunistic infection or neoplasm (including aerosolized or intravenous pentamidine) that develops during the study.

Concurrent Treatment:

Allowed:

* Any standard or experimental treatment for an opportunistic infection or neoplasm that develops during the study.

Patients must have AIDS with at least one cytologically or histologically proven episode of Pneumocystis carinii pneumonia (PCP).

* Patients must be free of acute medical problems.

Prior Medication:

Allowed:

* Zidovudine (AZT).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Requiring ongoing active therapy for an opportunistic infection at the time of study entry.
* Toxoplasmosis.
* Cryptococcus.
* Pulmonary Kaposi's sarcoma (KS).
* Asthma poorly controlled by medication.

Concurrent Medication:

Excluded:

* Pentamidine by any route other than aerosolized or intravenous or any other experimental agent for chemoprophylaxis of PCP while on the study (e.g.:
* Septra, Fansidar, Dapsone, or eflornithine).

Concurrent Treatment:

Excluded:

* Transfusion dependency defined as > 1 blood transfusion per month.

Patients with the following are excluded:

* Requiring ongoing active therapy for an opportunistic infection (O.I.) at the time of entry or having either Toxoplasmosis or cryptococcosis at entry.
* Pulmonary Kaposi's sarcoma (KS).
* Active substance abuse by patients who cannot comply with study procedures.
* Unwilling to sign informed consent.
* In the opinion of the investigator cannot cooperate with study procedure.
* Asthma poorly controlled by medication.
* Patients may not receive pentamidine by any other route than aerosolized or intravenous or any other experimental agent for chemoprophylaxis of PCP while on the study (e.g.:
* Septra, Fansidar, Dapsone, or eflornithine).

Prior Medication:

Excluded within 30 days of study entry:

* Antiretroviral agents, excluding zidovudine (AZT).
* Immunomodulating agents.
* Corticosteroids.

Prior Treatment:

Excluded within 7 days of study entry:

* Blood transfusion.
* Excluded:
* Requiring ongoing active treatments for an opportunistic infection at time of study entry.

Active substance abuse by patients who cannot comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Fisons Corp, Rochester, New York, United States